CLINICAL TRIAL: NCT05322187
Title: Sequential PD-1/PD-L1 Inhibitor and LENvatinib in Transitional Liver Cell Tumors（TLCT）and Refractory Hepatoblastoma for Young Adolescent and Pediatric Participants After Chemotherapy：a Cohort Study
Brief Title: Sequential PD-1/PD-L1 Inhibitor and LENvatinib in TLCT and Refractory Hepatoblastoma After Chemotherapy
Acronym: sPLENTY-pc
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RenJi-IIT2022-241
Record Dates: First submitted 2022-04-03; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Transitional Cell Tumor; Hepatoblastoma; Liver Cancer; Pediatric Solid Tumor; Pediatric Cancer
MeSH Terms: conditions — Hepatoblastoma; Liver Neoplasms; Neoplasms | interventions — Immune Checkpoint Inhibitors; lenvatinib; camrelizumab; pembrolizumab; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLEN(PD-1/PD-L1 inhibitor and LENvatinib) (Experimental): Treatment of PD-1/PD-L1 Inhibitor and LENvatinib would be employed in PLEN
  Interventions: Drug: PD-1 inhibitor

INTERVENTIONS:
Drug: PD-1 inhibitor — Sequential PD-1/PD-L1 Inhibitor and LENvatinib treatment after chemotherapy resistance
  Other Names: PD-L1 inhibitor; lenvatinib; Camrelizumab; Pembrolizumab; Duvarizumab; Sintilimab

SUMMARY:
This is a single arm, open-label trial studying the combination of PD-1/PD-L1 Inhibitor (e.g.pembrolizumab, Sintilimab,Duvarizumab，Camrelizumab )and lenvatinib given at the recommended dose in pediatric and young adolescent patients((5 year-old<age<14 year-old) with TLCT or refractory hepatoblastoma after chemotherapy.

DETAILED DESCRIPTION:
Transitional liver cell tumors exhibit an unusual phenotype with respect to clinical presentation, histopathology, immunohistochemistry, and treatment response. These apparently novel, unusual, and aggressive tumors occurring in older children and adolescents may form a transition in the putative developmental pathway of hepatocarcinogenesis, and usually refractory, resistant to chemotherapy.

The sPLENTY-pc is a perspective cohort study, investigating the efficiency of sequential combined usage of PD-1 Inhibitor (e.g.pembrolizumab, Sintilimab,Camrelizumab ) or PD-L1 inhibitor (Duvarizumab) plus lenvatinib given at the recommended dose in pediatric >5 year-old and young adult patients<14 yo with TLCT or refractory hepatoblastoma after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >= than 5 years and =< 14 years of age at the time of study enrollment
* pathological diagnosis of TLCT/NOS, or hepatoblastoma（HB）（Emergent Treatment for HB In emergency situation when a patient meets all other eligibility criteria and has had baseline required observations, but is too ill to undergo a biopsy safely, the patient may be enrolled without a biopsy.）
* Failed prior first-line or second-line chemotherapy
* general charactoristics: Lansky performance status 50-100% in patients ≤ 10 years of age OR Karnofsky performance status 50-100% in patients > 10 years of age Life expectancy > 8 weeks Hemoglobin > 8 g/dL Absolute neutrophil count > 1,000/mm^3 Platelet count > 100,000/mm^3 Total bilirubin ≤ 5 x upper limit of normal (ULN) for age, Aspartate aminotransferase (AST) or Alanine transaminase (ALT) < 10 x upper limit of normal (ULN) for age. Serum creatinine ≤ 3 times normal Normal metabolic parameters (i.e., serum electrolytes, glucose, calcium, and phosphate) Not pregnant or nursing No severe uncontrolled infection or enterocolitis
* Recovered from toxicity of prior therapy No chemotherapy within 3 weeks prior to study entry No prior PD1/PD-L1 blockade treatment

Exclusion Criteria:

* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.
* Patients who are currently receiving another investigational drug.
* Patients who are currently receiving other anticancer agents.
* Patients with uncontrolled infection.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of PD1/PD-L1 blockade

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2022-04-10 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (complete response/partial response) | up to 1 year
  Determined using Response Evaluation Criteria in Solid Tumors version 1.1. A responder is defined as a patient who achieves a best response of partial response or complete response on the study. Response rates will be calculated as the percent of evaluable patients who are responders, and confidence intervals will be constructed using the Wilson score interval method.
dynamic α-fetoprotein response (AFP-R) | up to 6 months for unresectable.
  The AFP-R was measured as the difference between maximum and final pre-liver transplant/resection AFP level, if surgery is not possible, the final level of AFP would be measured as the AFP at 6 month.

SECONDARY OUTCOMES:
Incidence and severity of study treatment-related adverse events measured by the Common Terminology Criteria for Adverse Events (CTCAE) v. 5 | up to 12 months
  oxicities will be defined using the Common Terminology Criteria for Adverse Events (CTCAE) v. 5.
Health outcomes as assessed by the PROMIS® Pediatric Scale v1.0 Global Health 7+2 scores at baseline, prior to start of each cycle, and last trial visit | up to 12 months
  Each question will be rated from the following: Excellent (5) to Poor (1), Never (5) to Always (1), or Never (1) to Almost Always (5)

CONTACTS AND LOCATIONS:
Overall Officials: Hao Feng, Principal Investigator — Dept. Liver Surgery, Renji Hospital, School of Medicine, SJTU; Qiang Xia, Study Chair — Dept. Liver Surgery, Renji Hospital, School of Medicine, SJTU
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China